CLINICAL TRIAL: NCT01038024
Title: A Pilot Study for the LC-MS/MS Assessment of Oxidative DNA Damage in Relation to Antioxidant Usage
Brief Title: Study for the Liquid Chromatography-mass Spectrometry (LC-MS/MS) Assessment of Oxidative DNA Damage in Relation to Antioxidant Usage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 155409
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Cancer
Keywords: antioxidant supplement
MeSH Terms: conditions — Neoplasms | interventions — Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antioxidant Supplements (Experimental)
  Interventions: Dietary Supplement: 1 tablet composed of antioxidants and minerals

INTERVENTIONS:
Dietary Supplement: 1 tablet composed of antioxidants and minerals — 1 tablet daily

SUMMARY:
The purpose of this study is to evaluate the basis for the reported good effects of antioxidant supplementation. A blood test using Mass Spectrometry will measure DNA damage which is expected to decrease with antioxidant administration and therefore decrease the risk of cancer.

DETAILED DESCRIPTION:
In this pilot study, the overall purpose is to establish the molecular basis for the hypothesis that oxidative stress is a risk factor for cancer. This will be achieved by establishing base line levels of oxidative DNA damage in a population of healthy individuals before and after taking antioxidant and mineral supplements for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Health male or female non-melanoma patients or volunteers
* 18 years or older with a life expectancy greater than 6 months
* Willing to provide pre and post blood samples to measure five DNA modifications in white blood cells
* Willing to participate in a one tablet a day eight week supplement program and to record the ingestion of the supplement on a participant calendar
* Must have never smoked or has not smoked for at least 6 months
* Informed of the investigational nature of the study, is able to provide informed consent and has signed thee informed consent form

Exclusion Criteria:

* Patients/healthy volunteers not meeting all of the above selection criteria.
* Patients/healthy volunteers who have a history of kidney stones within the last 5 years.
* Any participant with life threatening conditions including but not limited to cardiac failure, congestive heart failure, unstable coronary artery disease, uncontrolled hypertension, poorly controlled diabetes mellitus, kidney and liver disease,severe metabolic disorders and advanced cancer
* Patients not willing to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To establish a base line level for 5 DNA modifications of White blood cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Zeitouni, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States